CLINICAL TRIAL: NCT04057170
Title: Comparison of the Effects of Mulligan Mobilization With Movement Method and Accelerated Rehabilitation Protocol on Shoulder Pain and Functions in Subacromial Pain Syndrome: A Randomized Single Blind Trial
Brief Title: Manual Therapy Versus Conventional Rehabilitation Protocol on Subacromial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Volkan Deniz, PT, Director, Clinical Research, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Subacromial Impingement Syndrome
Keywords: shoulder pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mulligan method (Experimental): Mulligan mobilization with mowement method every three days for six weeks
  Interventions: Other: accelerated protocol and mulligan method
- accelerated protocol (Experimental): accelerated rehabilitation protocol every three days for six weeks
  Interventions: Other: accelerated protocol and mulligan method

INTERVENTIONS:
Other: accelerated protocol and mulligan method — manual therapy technic

SUMMARY:
This study compares the periodic effects of Accelerated rehabilitation protocol (ARP) and Mulligan mobilization with mowement method (MWM) in subacromial pain syndrome patients rehabilitation. Half of the participants will receive ARP, while the other half will receive MWM.

ELIGIBILITY:
Inclusion Criteria:

* to be in the 18-60 age range, to be cooperative during evaluation and treatment and to accept to participate in the study

Exclusion Criteria:

* the presence of adhesive capsulitis, surgical indication or shoulder surgery, cervicothoracic problems (such as stenosis and disc herniation) diagnosed as neurological or inflammatory joint diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index | two weeks
  It consists of 13 questions in two sections as 5 pain questions and 8 disability questions. Both sections are scored with VAS. The total score range is between 0-130 and it is calculated with the percentage score. Pain and disability are inversely proportional with the percentage score
Visual Analogue Scale | two weeks
  to record pain intensity during rest and active shoulder movements. The patient is asked to mark the point corresponding to the pain (0 no pain and 10 maximal pain) on 10 cm horizontal line. The distance between the marked point and the beginning is recorded as a pain score
Active Range of Motion measurement | two weeks
  Conventional goniometer with 1° increments is used to determine shoulder limitations due to pain in patients
Subacromial Interval Measurement | six weeks
  Subacromial interval measurement was performed via anterior-posterior shoulder radiography

CONTACTS AND LOCATIONS:
Locations (1):
- Volkan Deniz, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No